CLINICAL TRIAL: NCT02402868
Title: Intranasal Ketamine Versus Intravenous Ketamine for Procedural Conscious Sedation in Children: a Multi-centre Randomized Controlled Non-inferiority Trial
Brief Title: Intranasal Versus Intravenous Ketamine for Procedural Sedation in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Naveen Poonai, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106549
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Bone Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal ketamine and saline (Experimental): Intranasal ketamine (each single dose, 8 mg/kg prepared in 0.9% NS in 3 mL syringe and atomizer, to a maximum of 6.4 mL) PLUS IV 0.9% NS 0.02 mL/kg
  Interventions: Drug: Ketamine and saline
- Intravenous ketamine and saline (Active Comparator): Intravenous ketamine (single dose, 1 mg/kg, to a maximum 100 mg) PLUS intranasal 0.9% NS 0.08 mL/kg divided to both nares
  Interventions: Drug: Ketamine and saline

INTERVENTIONS:
Drug: Ketamine and saline — Ketamine intravenous and intranasal
  Other Names: Ketamine hydrochloride

SUMMARY:
This study will examine the effectiveness of intranasal (IN) ketamine compared to standard intravenous (IV) ketamine administration for simple reductions of orthopaedic injuries in the paediatric population. The aim is to assess if IN administration is equivalent to the current standard of care, IV. The population to be studied is children 5-17 years of age who require a simple orthopaedic reduction. Following a double dummy approach to overcome the difficulty in masking interventions, each participant will recieve both IV and IN interventions, only one of which will be the real drug. Procedural conscious sedation (PCS) will be assessed using the University of Michigan Sedation Scale (UMSS).

DETAILED DESCRIPTION:
Randomization and concealment of allocation will be pharmacy-controlled using a computer-based random number generator. The treating physician, research assistant, and participant will be blinded to the intervention. Eligible participants will be randomized in a 1:1 allocation ratio with a stratified block design of six to either (1) IN ketamine (each single dose, 8 mg/kg prepared in 0.9% NS in 3 mL syringe and atomizer, to a maximum of 1.5 mL) PLUS IV 0.9% NS 0.02 mL/kg or (2) IV ketamine (single dose, 1 mg/kg, to a maximum 100 mg) PLUS intranasal 0.9% NS 0.08 mL/kg divided to both nares. Due to the perceptible differences in interventional routes, each participant will receive both IV and IN interventions using this double-dummy approach. For IN dose volumes less than or equal to 0.5 mL, the entire dose will be delivered into 1 nostril and for doses greater than 0.5 mL, the dose will be divided equally between both nares. Adjuctive sedation will be given as needed in the form of IV ketamine, 1 mg/kg every 10 minutes for participants who do not achieve adequate sedation at 20 minutes (UMSS score of 4). A figure of the atomizer device used to deliver the IN agent has been uploaded. Eligible participants (defined in section 2.5 above) will be identified by the treating physician after viewing the radiographs and performing a clinical assessment. The physician will then inform a research assistant (RA) that the participant is eligible. The RA will then seek informed consent and explain the protocol to the family. Baseline demographic information will be obtained. Informed consent for PCS and a pre-anesthetic assessment will be performed by the treating physician in accordance with the usual standard of care. UMSS scores will be obtained by a trained RA at 5 minutes pre-intervention, intervention (0 minutes) and every 5 minutes thereafter for 60 minutes post-intervention or until the participant is ambulatory and drinking well, whichever is longer. Participants will receive standard monitoring of oxygen saturation, blood pressure, respiratory rate, apnea, heart rate, and rash by the attending nurse and physician every 5 minutes as per the usual standard of care. The usual standard of care also includes monitoring post-anesthetic for the presence of known idiosyncratic effects of ketamine that include vomiting, seizure, headache, emergence reaction, and hypersensitivity. The RA will obtain this information from the nursing record at discharge. Immediately prior to discharge, the RA will also record the duration of stay in the ED and parental satisfaction with PCS. 1. Chiaretti et al. 2011. Intranasal lidocaine and midazolam for procedural sedation in children. Arch Dis Child. 96;160-163

ELIGIBILITY:
Inclusion Criteria:

* Patients 5-17 years (up to 80 kg) presenting to the paediatric ED who require a PCS for an acute simple orthopedic injuries who require a procedural sedation and analgesia (PSA). A "simple" injury is defined as a fracture or dislocation that: 1) Angulated with or without displacement but is not shortened) 2) Non-comminuted

Exclusion Criteria:

* 1) Previous hypersensitivity reaction to ketamine including rash, difficulty breathing, hypotension, apnea, or laryngospasm 2) Globe rupture 3) Traumatic brain injury with intracranial hemorrhage 4) History of uncontrolled hypertension 5) Nasal bone deformity 6) Fracture reduction expected to require > 20 minutes 7) Poor English fluency 8) American Society of Anesthesiologists (ASA) class of 3 or greater 9) Previous sedation with ketamine within 24 hours of index visit 10) Known diagnosis of schizophrenia or active psychosis 11) Pregnancy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
University of Michigan Sedation Score | From the time the IV intervention is given to 60 minutes post intervention or when drinking, whichever is longer
  The primary outcome is the UMSS score at 10 minutes post administration of the IV intervention compared to UMSS score immediately prior to the first IN intervention (delta) using the University of Michigan Sedation Scale (UMSS)

SECONDARY OUTCOMES:
Onset of sedation | Within 1 hour following intervention
  Time interval from first IN spray to UMSS score of greater than 3 in minutes
Duration of sedation | Within 2 hours following sedation
  Time interval from UMSS score greater than 3 to a UMSS score of 0 in minutes
Adverse events | Within 2 hours following sedation
  Obtained when patient fully awake and prior to discharge from the participant, physician report and corroborated with nursing sedation record
Length of stay | Within 3 hours of intervention
  Time from arrival in ED bed to discharge in minutes
Length of stay due to sedation | Within 3 hours of intervention
  Time from first IN spray to discharge in minutes
Duration of procedure | Within 3 hours of intervention
  Time from first IN spray to end of cast application
Parental satisfaction | Within 2 hours of sedation
  Obtained immediately prior to discharge using a 5-item Likert scale; Parents not wishing to remain in proximity of child for sedation may opt out
Child satisfaction | Within 2 hours of sedation
  Obtained immediately prior to discharge using a 5-item Likert scale
Sedating physician satisfaction | Duration of ED visit
  Obtained immediately prior to discharge using a 5-item Likert scale
Adjunctive sedative medication | Duration of ED visit
  Number of doses and type of adjunctive sedative medication required
Analgesic medication | Duration of ED visit
  Number of doses and type of analgesic medication required
Pain | 15 minutes prior to and 2 hours post intervention
  Child's self reported pain score using the Faces Pain Scale - Revised
Emergence Agitation | Every 5 minutes for 60 minutes starting 20 minutes post IV intervention
  Degree of emergency agitation and delirium as recorded by observer using the Paediatric Anesthesia Emergency Delirium (PAED) scale
Nasal Irritation | Within 1 hour of intervention
  Recorded using a 5-item Likert scale anchored from 1=none to 5=very severe when child has a UMSS score of 0 and is awake and drinking
Successful sedation | From time of first IN spray to when participant is fully awake (UMSS score of 0 for 15 minutes)
  Successful sedation - Based on the definition of Bhatt et al., this will be defined as no unpleasant patient recall of the procedure, no resistance or restraint required during the procedure, no permanent sedation-related complication or no sedation-related event requiring abandonment of the procedure.
  Defined as: no unpleasant patient recall of the procedure, no resistance or restraint required during the procedure, no permanent sedation-related complication or no sedation-related event requiring abandonment of the procedure.
  Defined as no unpleasant recall of procedure, no resistance or restraint, no permanent sedation related complication, no sedation-related event requiring abandonment of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, Principal Investigator — Western University
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No